CLINICAL TRIAL: NCT00753324
Title: Routine Use of Antiretroviral Therapy to Prevent Mother-to-Child HIV Transmission in the Kafue District of Zambia (Impact of HAART to Prevent Pediatric AIDS in Rural Zambia).
Brief Title: Routine Use of Antiretroviral Therapy to Prevent Mother-to-Child HIV Transmission in the Kafue District of Zambia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Principal Investigator, Benjamin Chi, MD, MSc, Associate Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CIDRZ 1222/F070821006
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: HIV Infections
Keywords: PMTCT; HAART; Pregnancy; HIV Infection; HIV Transmission; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine three-drug antiretroviral prophyalxis (Experimental): Cohort of 160 HIV-infected women, approached at > 28 weeks gestation and initiated on routine HAART for the purposes of PMTCT.
  Interventions: Drug: Routine three-drug antiretroviral prophylaxis
- Control arm (No Intervention): A cohort of 160 women will be enrolled from the control clinics, from 28 weeks gestation onward. At these sites, the antenatal zidovudine will be offered, with provision of single-dose nevirapine for self-administration in labor. This practice is in accordance with the current standard of care recommended by the Zambian National Guidelines for PMTCT.

INTERVENTIONS:
Drug: Routine three-drug antiretroviral prophylaxis — Women who are identified as HIV-infected will be offered routine combination antiretroviral prophylaxis starting at 28 weeks gestation (timing consistent with Zambian national guidelines for short-course ZDV). The first-line combination provided to pregnant women will be standardized following consultation with the Ministry of Health, but will likely include ZDV, lamivudine (3TC) and either NVP or lopinavir / ritonavir. In women who with moderate to severe anemia, ZDV is substituted with stavudine (d4T). In accordance with the Zambian national guidelines, any patients who are started on NVP will begin with a once daily dose for two weeks before increasing to the regular twice daily schedule
  Arms: Routine three-drug antiretroviral prophyalxis

SUMMARY:
The investigators will enroll a cohort of HIV-infected pregnant women accessing PMTCT services, to better understand the incremental benefits (e.g. reduction in HIV transmission, improvements in HIV-free survival) and risks (e.g. drug toxicities) of the routine HAART strategy, in comparison to HIV-infected pregnant women accessing the Zambian Standard of Care services.

The investigators will test the hypothesis that routine use of HAART produces significant reductions in HIV transmission rates, with only minimal side effects.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* Pregnant women
* Ability to provide informed consent.
* Meets eligibility criteria for HAART initiation

Exclusion Criteria:

* Unwillingness to provide informed consent
* Below the age of legal consent

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2009-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
HIV Infection | 12 months

SECONDARY OUTCOMES:
HIV Infection | 6 weeks, 6 months and 24 months
Infant survival | 12 and 24 months
HIV-free survival | 12 months and 24 months
Incidence of maternal toxicity to HAART regimens | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Chi, M.D, Principal Investigator — Centre for Infectious Disease Research in Zambia
Locations (1):
- CIDRZ, Lusaka, Lusaka Province, Zambia

REFERENCES:
- [Result] Gartland MG, Chintu NT, Li MS, Lembalemba MK, Mulenga SN, Bweupe M, Musonda P, Stringer EM, Stringer JS, Chi BH. Field effectiveness of combination antiretroviral prophylaxis for the prevention of mother-to-child HIV transmission in rural Zambia. AIDS. 2013 May 15;27(8):1253-62. doi: 10.1097/QAD.0b013e32835e3937. PMID 23324656